CLINICAL TRIAL: NCT01436474
Title: The Role of Varenicline in Treating Opioid Dependence: A Pilot Study
Brief Title: Pilot Study of Varenicline to Treat Opioid Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, W. Michael Hooten, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-002062
Record Dates: First submitted 2011-06-03; First posted 2011-09-19 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Pain; Opioid Dependence
Keywords: Varenicline; Chantix; Chronic Pain; Opioid dependence
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental): We will be comparing Varenicline to placebo in a single-blinded placebo controlled, randomized study
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): We will be using a placebo in a randomized, controlled, single-blinded trial to look at varenicline for the indication of facilitating opioid tapering in opioid-dependent patients with chronic pain.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Patients will be randomly assigned to receive either varenicline or placebo for 45 days. Patients assigned to varenicline and are current smokers will receive 0.5mg by the oral route once a day for 3 days, followed by 0.5mg twice a day for 4 days. After the first week the dose will be increased to 1mg twice daily for the remainder of the active treatment period of the study. Patients assigned to varenicline and are non-smokers will receive 0.5mg by the oral route once a day for 6 days, followed by 0.5mg twice a day for 6 days. After the first 12 days the dose will be increased to 1mg twice daily for the remainder of the active treatment period of the study. Patients assigned to placebo will receive identical looking capsules in a dosage schedule similar to varenicline.
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Patients will be randomly assigned to receive either varenicline or placebo for 45 days. Patients assigned to varenicline and are current smokers will receive 0.5mg by the oral route once a day for 3 days, followed by 0.5mg twice a day for 4 days. After the first week the dose will be increased to 1mg twice daily for the remainder of the active treatment period of the study. Patients assigned to varenicline and are non-smokers will receive 0.5mg by the oral route once a day for 6 days, followed by 0.5mg twice a day for 6 days. After the first 12 days the dose will be increased to 1mg twice daily for the remainder of the active treatment period of the study. Patients assigned to placebo will receive identical looking capsules in a dosage schedule similar to varenicline.
  Other Names: chantix
  Arms: Placebo

SUMMARY:
The objective of this proposal is to explore the potential of varenicline as a pharmacotherapeutic agent for opioid dependence and addiction.

ELIGIBILITY:
Inclusion criteria

* Age>=21 years
* Use of opioids at admission to PRC, with daily morphine equivalent dose>=60mg
* Be able and willing to participate fully in all aspects of the study including one month follow-up after completion of PRC
* Ability to provide informed consent

Exclusion criteria

* Currently using varenicline or other pharmacotherapy for nicotine dependence
* Currently pregnant, lactating, or likely to become pregnant during the trial and not willing to use an acceptable form of contraception;
* History of a major cardiovascular event in the past 6 months including unstable angina, acute myocardial infarction, stroke, or coronary angioplasty;
* Known varenicline allergy
* Use of any medication (e.g., methadone, Suboxone) as maintenance therapy for opiate addiction
* Identification of illicit drugs (e.g., marijuana, cocaine) on the baseline urine toxicology screen

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
assessment of opioid withdrawal symptoms | 45 days
  During their treatment, patients are closely monitored by a multidisciplinary team, and there are regular assessments of pain, depression, substance use, and pain-related physical and emotional functioning
Assessment of cravings at one month following opioid tapering | 45 days
  During their treatment, patients are closely monitored by a multidisciplinary team, and there are regular assessments of pain, depression, substance use, and pain-related physical and emotional functioning

CONTACTS AND LOCATIONS:
Overall Officials: William Hooten, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States